CLINICAL TRIAL: NCT02940379
Title: A Two-cohort, Open-label, Fixed-sequence, Two-period, Two-treatment Pharmacokinetic Interaction Study of Repeated Oral Doses of Sotagliflozin on a Single Dose Cocktail of Metoprolol and Midazolam Used as Probe Substrates for CYP2D6 and CYP3A Activities, Respectively, in Healthy Subjects
Brief Title: A Drug to Drug Interaction Study of Sotagliflozin With Midazolam and Metoprolol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT14972; U1111-1184-8677 (Other: UTN)
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Midazolam; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Participants will initially be given with treatment A (cocktail of metoprolol and midazolam) and then will start with treatment B (Dose 1 of Sotagliflozin plus cocktail) after 3 days
  Interventions: Drug: sotagliflozin (SAR439954); Drug: midazolam; Drug: metoprolol
- Cohort 2 (Experimental): Participants will initially be given with treatment A (cocktail of metoprolol and midazolam) and then will start with treatment B (Dose 2 of Sotagliflozin plus cocktail) after 3 days
  Interventions: Drug: sotagliflozin (SAR439954); Drug: midazolam; Drug: metoprolol

INTERVENTIONS:
Drug: sotagliflozin (SAR439954) — Pharmaceutical form: tablet
  Route of administration: oral
Drug: midazolam — Pharmaceutical form: HCl syrup
  Route of administration: oral
Drug: metoprolol — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To assess the effect of repeated once-daily oral doses of sotagliflozin on CYP2D6 and CYP3A activities using a CYP probe cocktail of metoprolol and midazolam.

Secondary Objective:

To assess the clinical and laboratory safety of sotagliflozin coadministered with the cocktail probes as compared to that of cocktail probes alone.

DETAILED DESCRIPTION:
The total study duration per subject is up to 58 days.

ELIGIBILITY:
Inclusion criteria :

* Male or female healthy subjects, between 18 and 55 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 30.0 kg/m^2, inclusive.
* Normal vital signs, electrocardiogram (ECG), and laboratory parameters
* Female subjects must use a double contraception method during the study, except if she has undergone sterilization at least 3 months earlier or is postmenopausal. The accepted double contraception methods include the use of one of the following contraceptive options: (1) condom; (2) diaphragm or cervical/vault cap; (3) spermicide in addition to the use of one of the following: a) Intrauterine device (IUD); b) Vasectomized partner; c) Sexual abstinence. Hormonal contraception is NOT acceptable in this study.

Exclusion criteria:

Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.

Frequent headaches and/or migraine, recurrent nausea and/or vomiting.

* Blood donation, any volume, within 2 months before inclusion.
* Symptomatic postural hypotension.
* Presence or history of drug hypersensitivity, allergic disease or asthma diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse.
* If female, pregnancy or breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion. Any oral contraceptives during the screening period or for at least 15 days prior to the first dose of Period 1; any injectable contraceptives or hormonal intrauterine devices within 12 months prior to the first dose of Period 1; or topical controlled delivery contraceptives (patch) for 3 months prior to the first dose of Period 1.
* Any contra-indications to metoprolol, according to the applicable labeling.
* Any contra-indications to midazolam, according to the applicable labeling.
* Any consumption of citrus (grapefruit, orange, etc.) or their juices within 5 days before inclusion.
* Any history or presence of deep leg vein thrombosis or embolism or a recurrent or frequent appearance of deep leg vein thrombosis in first degree relatives (parents, siblings or children).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assessment of midazolam pharmacokinetic (PK) parameter: Area under the curve (AUC) | Day 1 to Day 2 of Treatment A Period
Assessment of midazolam PK parameter: AUC | Day 11 to Day 12 of Treatment B Period
Assessment of metoprolol PK parameter: AUC | Day 1 to Day 3 of Treatment A Period
Assessment of metoprolol PK parameter: AUC | Day 11 to Day 13 of Treatment B Period

SECONDARY OUTCOMES:
Assessment of PK parameter: maximum plasma concentration (Cmax) | Day 1 to Day 2 of Treatment A Period (midazolam)
Assessment of PK parameter: Cmax | Day 11 to Day 12 of Treatment B Period (midazolam)
Assessment of PK parameter: Cmax | Day 1 to Day 3 of Treatment A Period (metoprolol)
Assessment of PK parameter: Cmax | Day 11 to Day 13 of Treatment B Period (metoprolol)
Assessment of PK parameter: time to reach Cmax (Tmax) | Day 1 to Day 2 of Treatment A Period (midazolam)
Assessment of PK parameter: Tmax | Day 11 to Day 12 of Treatment B Period (midazolam)
Assessment of PK parameter: Tmax | Day 1 to Day 3 of Treatment A Period (metoprolol)
Assessment of PK parameter: Tmax | Day 11 to Day 13 of Treatment B Period (metoprolol)
Assessment of PK parameter: terminal-half life (t1/2z) | Day 1 to Day 2 of Treatment A Period (midazolam)
Assessment of PK parameter: t1/2z | Day 11 to Day 12 of Treatment B Period (midazolam)
Assessment of PK parameter: t1/2z | Day 1 to Day 3 of Treatment A Period (metoprolol)
Assessment of PK parameter: t1/2z | Day 11 to Day 13 of Treatment B Period (metoprolol)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 840001, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org